CLINICAL TRIAL: NCT05361720
Title: Optimal Treatment by Invoking Biologic Clusters in Renal Cell Carcinoma (OPTIC RCC)
Brief Title: Genetic Testing to Select Therapy for the Treatment of Advanced or Metastatic Kidney Cancer, OPTIC RCC Study
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Vanderbilt-Ingram Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH); United States Department of Defense (U.S. Federal Agency)
Responsible Party: Principal Investigator, Brian Rini, Principal Investigator, Vanderbilt-Ingram Cancer Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VICCURO21103; NCI-2022-03150 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); VICCURO21103 (Other: Vanderbilt University/Ingram Cancer Center); P30CA068485 (NIH); CDMRP-KC210255 (Other: Department of Defense)
Record Dates: First submitted 2022-04-25; First posted 2022-05-05 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Advanced Clear Cell Renal Cell Carcinoma; Metastatic Clear Cell Renal Cell Carcinoma; Stage III Renal Cell Cancer AJCC v8; Stage IV Renal Cell Cancer AJCC v8
MeSH Terms: conditions — Clear-cell metastatic renal cell carcinoma; Carcinoma, Renal Cell | interventions — cabozantinib; Ipilimumab; CTLA-4 Antigen; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm I (ipilimumab, nivolumab) (Experimental): INDUCTION: Patients receive ipilimumab and nivolumab IV on day 1. Cycles repeat every 21 days for 4 cycles.
  MAINTENANCE: Patients receive nivolumab IV on day 1. Cycles repeat every 4 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Ipilimumab; Biological: Nivolumab
- Arm II (nivolumab, cabozantinib) (Experimental): Patients receive nivolumab IV on day 1 and cabozantinib PO QD. Cycles repeat every 4 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Cabozantinib; Biological: Nivolumab

INTERVENTIONS:
Drug: Cabozantinib — Given PO
  Arms: Arm II (nivolumab, cabozantinib)
Biological: Ipilimumab — Given IV
  Other Names: Anti-Cytotoxic T-Lymphocyte-Associated Antigen-4 Monoclonal Antibody; BMS-734016; Ipilimumab Biosimilar CS1002; MDX-010; MDX-CTLA4; Yervoy
  Arms: Arm I (ipilimumab, nivolumab)
Biological: Nivolumab — Given IV
  Other Names: BMS-936558; CMAB819; MDX-1106; NIVO; Nivolumab Biosimilar CMAB819; ONO-4538; Opdivo

SUMMARY:
This phase II trial tests whether using genetic testing of tumor tissue to select the optimal treatment regimen works in treating patients with clear cell renal cell (kidney) cancer that has spread to other places in the body (advanced or metastatic). The current Food and Drug Administration (FDA)-approved regimens for advanced kidney cancer fall into two categories. One treatment combination includes two immunotherapy drugs (nivolumab plus ipilimumab), which are delivered by separate intravenous infusions into a vein. The other combination is one immunotherapy drug (nivolumab infusion) plus an oral pill taken by mouth (cabozantinib). Nivolumab and ipilimumab are "immunotherapies" which release the brakes of the immune system, thus allowing the patient's own immune system to better kill cancer cells. Cabozantinib is a "targeted therapy" specifically designed to block certain biological mechanisms needed for growth of cancer cells. In kidney cancer, cabozantinib blocks a tumor's blood supply. The genetic (DNA) makeup of the tumor may affect how well it responds to therapy. Testing the makeup (genes) of the tumor, may help match a treatment (from one of the above two treatment options) to the specific cancer and increase the chance that the disease will respond to treatment. The purpose of this study is to learn if genetic testing of tumor tissue may help doctors select the optimal treatment regimen to which advanced kidney cancer is more likely to respond.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To improve objective response rate of front-line therapy in advanced renal cell carcinoma (RCC) by prospectively assigning ipilimumab/nivolumab or nivolumab/cabozantinib according to a patient's ribonucleic acid sequence (RNAseq)-defined biologic cluster.

SECONDARY OBJECTIVE:

I. To assess clinical outcome of cluster-assigned treatment in front-line metastatic renal cell carcinoma (mRCC).

EXPLORATORY OBJECTIVE:

I. To assess tissue and peripheral blood for pharmacodynamic correlations with response to treatment.

OUTLINE: Patients are assigned to 1 of 2 arms.

ARM I:

INDUCTION: Patients receive ipilimumab and nivolumab intravenously (IV) on day 1. Cycles repeat every 21 days for 4 cycles.

MAINTENANCE: Patients receive nivolumab IV on day 1. Cycles repeat every 4 weeks in the absence of disease progression or unacceptable toxicity.

ARM II: Patients receive nivolumab IV on day 1 and cabozantinib orally (PO) once a day (QD). Cycles repeat every 4 weeks in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up within 30 days from last dose.

ELIGIBILITY:
Inclusion Criteria:

* Histological confirmation of RCC with a clear cell component
* Advanced (not amenable to curative surgery or radiation therapy) or metastatic (American Joint Committee on Cancer [AJCC] stage IV) RCC
* Patient can comprehend and sign the study informed consent form
* Male or female >= 18 years of age at the time of informed consent
* Karnofsky performance status (KPS) of >= 70%
* No prior systemic therapy for RCC in the neoadjuvant, adjuvant or metastatic setting
* At least one measurable lesion as defined by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1
* Tumor tissue for ribonucleic acid (RNA)-sequencing (tumor tissue from bony metastasis is not suitable but a soft tissue component around bone is acceptable)

  * Screening tissue consent- Patient must be assigned to either Cluster 1/2 or 4/5. Patients assigned to cluster 3/6/7 will not be eligible for the treatment study
* Adequate renal function defined as calculated creatinine clearance >= 30 mL/min per the Cockcroft and Gault formula
* Adequate liver function defined by:

  * Total bilirubin =< 1.5 times the upper limit of normal (ULN) except for unconjugated hyperbilirubinemia of Gilbert's syndrome
  * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) =< 3 x ULN
* Women of childbearing potential (WOCBP) must have a negative serum pregnancy test during screening and prior to receiving first dose of protocol-indicated treatment

  * Women of childbearing potential (WOCBP) is defined as any female who has experienced menarche who has not undergone surgical sterilization (hysterectomy or bilateral oophorectomy) or is not postmenopausal
  * Menopause is defined clinically as 12 months of amenorrhea in a woman over 45 years of age in the absence of other biological or physiological causes

Exclusion Criteria:

* =< 14 days before first dose of protocol-indicated treatment:

  * Major surgery requiring general anesthesia
* Inadequately controlled hypertension (systolic blood pressure [SBP] > 160/90 mmHg)

  * Anti-hypertensive medications are permitted.
* Active infection requiring infusional treatment
* Has preexisting gastrointestinal or non-gastrointestinal fistula
* Proteinuria > 2 g/ 24 hours (hrs)

  * If patient has 1+ protein on urine dipstick then a 24 hr urine collection is required
* Non-healing wounds on any part of the body (for patients assigned to Cabo/Nivo only)
* Known clinically significant active bleeding including hemoptysis
* Inability to swallow oral medication; or the presence of a poorly controlled gastrointestinal disorder that could significantly affect the absorption of oral study drug (for patients assigned to Cabo/Nivo only) - e.g., Crohn's disease, ulcerative colitis, chronic diarrhea (defined as > 4 loose stools per day), malabsorption, or bowel obstruction
* Significant cardiovascular disease or condition including:

  * Class III or IV cardiovascular disease according to the New York Heart Association (NYHA) functional criteria
  * Unstable angina pectoris (i.e., last episode =< 3 months prior to first dose of protocol-indicated treatment)
  * Myocardial infarction within 3 months prior to starting treatment
* Subjects with central nervous system (CNS) metastases are eligible after they have completed local therapy (e.g., whole brain radiation therapy [WBRT], surgery or radiosurgery)
* Any condition requiring systemic treatment with either systemic corticosteroids (> 10 mg/day prednisone or equivalent daily) or other immunosuppressive medications within 14 days prior to initiating protocol-indicated treatment
* In the absence of active autoimmune disease: Subjects are permitted the use of corticosteroids with minimal systemic absorption (e.g., topical, ocular, intra-articular, intranasal, and inhalational), =< 10 mg/day prednisone or equivalent daily; and physiologic replacement doses of systemic corticosteroids =< 10 mg/day prednisone or equivalent daily (e.g., hormone replacement therapy needed in patients with hypophysitis)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2022-12-01 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Overall response rate (ORR) (Arm 1) | Up to 4 years
  Assessed per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1. ORR = complete response (CR) + partial response (PR). The Agresti-Coull two-sided 95% confidence intervals (CIs) for the success rate will be reported.
Overall response rate (Arm 2) | Up to 4 years
  Assessed per RECIST 1.1. ORR = CR + PR. The Agresti-Coull two-sided 95% CIs for the success rate will be reported.

SECONDARY OUTCOMES:
Progression free survival | Up to 4 years
  Possible risk factors will be compared for survival with Kaplan-Meier estimates and log-rank tests. The proportional hazards model will be used for adjusting tests of significance and estimating the hazard ratios. Will apply the generalized estimating equation (GEE) statistical procedure for longitudinal binary data analysis with multiple observable vectors for the same subject. For the continuous multiple time points or correlated data, will use the mixed effects model to conduct the profile analysis. The adjusted 95% CIs will be reported.
Depth of response > 80% | At 6 months
  Will apply the GEE statistical procedure for longitudinal binary data analysis with multiple observable vectors for the same subject. For the continuous multiple time points or correlated data, will use the mixed effects model to conduct the profile analysis. The adjusted 95% CIs will be reported.
Incidence of immune-related adverse events | Up to 4 years
  Adverse medical events will be tabulated. National Cancer Institute toxicity grade 3 and grade 4 laboratory abnormalities will be listed.

CONTACTS AND LOCATIONS:
Overall Officials: Brian I Rini, MD, Principal Investigator — Vanderbilt University/Ingram Cancer Center
Locations (6):
- United States (6):
  - City of Hope National Medical Center, Duarte, California
  - Chao Family Comprehensive Cancer Center, Orange, California
  - University Hospitals Seidman Cancer Center, Cleveland, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - University of Texas, Southwestern Medical Center, Dallas, Texas

DOCUMENTS (1):
  • Informed Consent Form (2023-12-27): https://cdn.clinicaltrials.gov/large-docs/20/NCT05361720/ICF_000.pdf